CLINICAL TRIAL: NCT00320788
Title: A Randomized, Controlled Study of the Safety, Tolerability and Biological Effect of Repeated Intravitreal Administration of VEGF Trap in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Safety and Efficacy of Repeated Intravitreal Administration of Vascular Endothelial Growth Factor (VEGF) Trap in Patients With Wet Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGFT-OD-0508
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2012-03-01 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-01

CONDITIONS: Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- aflibercept injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q4 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)
- aflibercept injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q12 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)
- aflibercept injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q4 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)
- aflibercept injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q12 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)
- aflibercept injection (VEGF Trap-Eye, BAY86-5321) 4.0mg q12 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received 0.5 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 4 week intervals through Week 12
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q4
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received 0.5 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 12 week intervals through Week 12.
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q12
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received 2.0 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 4 week intervals through Week 12
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q4
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received 2.0 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 12 week intervals through Week 12.
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q12
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received 4.0 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 12 week intervals through Week 12.
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection (VEGF Trap-Eye, BAY86-5321) 4.0mg q12

SUMMARY:
This study examines the effect of intravitreally administered VEGF Trap in patients with wet AMD.

The purpose of this trial is to assess the ocular and systemic safety and tolerability of repeated intravitreal doses of VEGF Trap in patients with subfoveal choroidal neovascularization (CNV) due to AMD.

DETAILED DESCRIPTION:
This is a double masked, prospective, randomized study in which five groups of approximately 30 patients meeting the eligibility criteria will be randomly assigned in a balanced ratio to receive a series of intravitreal (IVT) injections of VEGF Trap into the study eye at 4- or 12 -week intervals over a 12-week period.

After Week 12, patients will be evaluated every 4 weeks. Patients will remain on study or may be eligible to enter a long-term extension study, in which they will continue to receive VEGF Trap.

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal CNV secondary to AMD.
* Central retinal (including lesion) thickness ≥ 300 µm as measured by Optical Coherence Tomography (OCT).
* Early Treatment of Diabetic Retinopathy Study (ETDRS) best-corrected visual acuity of 73 letters to 34 letters.

Exclusion Criteria:

* History of any vitreous hemorrhage within 4 weeks prior to Day 1.
* Aphakia.
* Significant subfoveal atrophy or scarring.
* Prior treatment with the following in the study eye:

  * Subfoveal thermal laser therapy.
  * Submacular surgery or other surgical intervention for the treatment of AMD.
  * Extrafoveal laser coagulation treatment within 12 weeks prior to Day 1.
  * Photodynamic therapy (PDT) within 12 weeks prior to Visit 2 (Day 1).
  * Pegaptanib sodium (Macugen) within 8 weeks of Visit 2 (Day 1).
  * Juxtascleral steroids or anecortave acetate within 24 weeks (6 months) prior to Visit 2 (Day 1).
  * Intravitreal administration of triamcinolone acetonide or other steroids within 24 weeks prior to Visit 2 (Day 1), unless no visible residue of drug substance can be seen in the vitreous cavity using indirect ophthalmoscopy.
  * Prior systemic or intravitreal treatment with VEGF Trap, ranibizumab (Lucentis) or bevacizumab (Avastin).
* Presence of any other condition or laboratory abnormality, which, in the opinion of the Investigator, would interfere with the assessment of disease status/progression or jeopardize the patient's appropriate participation in this Phase II study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (18):
- United States (18):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Centers, PC, Tucson, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Loma Linda University Health Care, Loma Linda, California
  - Southeast Retina Center, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Johns Hopkins Hospital School of Medicine, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants PC, West Springfield, Massachusetts
  - Charlotte Eye, Ear, Nose & Throat Asssociates, Charlotte, North Carolina
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest PC, Portland, Oregon
  - Retina Diagnostic and Treatment Assoc., LLC, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina-Vitreous Associates, P.C., Nashville, Tennessee
  - Vitreoretinal Consultants Scurlock Tower Texas Medical Center, Houston, Texas
  - Medical Center Ophthamology, San Antonio, Texas

REFERENCES:
- [Derived] Li E, Donati S, Lindsley KB, Krzystolik MG, Virgili G. Treatment regimens for administration of anti-vascular endothelial growth factor agents for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 May 5;5(5):CD012208. doi: 10.1002/14651858.CD012208.pub2. PMID 32374423
- See also: Primary endpoint results of a phase II study of vascular endothelial growth factor trap-eye in wet age-related macular degeneration. — http://www.ncbi.nlm.nih.gov/pubmed/21640257
- See also: The 1-year results of CLEAR-IT 2, a phase 2 study of vascular endothelial growth factor trap-eye dosed as-needed after 12-week fixed dosing. — http://www.ncbi.nlm.nih.gov/pubmed/21640258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 29 study sites in the United States. Recruitment period: May 2006 to April 2007.
Pre-assignment Details: A total of 301 participants were screened; 159 participants were randomized; 157 participants were included in both the Safety Analysis Set (SAF) and the Full Analysis Set (FAS) as all received study treatment, had baseline assessments and at least 1 post-baseline assessment.
Groups:
- Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q4: Participants received 0.5 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 4 week intervals through Week 12.
- Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q12: Participants received 0.5 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 12 week intervals through Week 12.
- Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q4: Participants received 2.0 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 4 week intervals through Week 12.
- Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q12: Participants received 2.0 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 12 week intervals through Week 12.
- Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 4.0mg q12: Participants received 4.0 mg of aflibercept injection (VEGF Trap-Eye, BAY86-5321) at 12 week intervals through Week 12.
Period: Overall Study
Arm/Group | Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q4 | Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 0.5mg q12 | Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q4 | Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 2.0mg q12 | Aflibercept Injection (VEGF Trap-Eye, BAY86-5321) 4.0mg q12
Started | 32 | 32 | 32 | 32 (Participants Randomized) | 31
Participants Received Treatment (SAF) | 32 | 32 | 31 (One participant in this group did not receive treatment and was not included in the SAF and FAS) | 31 (One participant in this group did not receive treatment and was not included in the SAF and FAS) | 31
Completed | 26 | 26 | 29 | 27 | 26
Not Completed | 6 | 6 | 3 | 5 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 0
Not completed — Decision by the Sponsor | 1 | 1 | 0 | 0 | 1
Not completed — Other | 1 | 2 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aflibercept Injection 0.5mg q4: Participants received 0.5 mg of aflibercept injection at 4 week intervals through Week 12.
- Aflibercept Injection 0.5mg q12: Participants received 0.5 mg of aflibercept injection at 12 week intervals through Week 12.
- Aflibercept Injection 2.0mg q4: Participants received 2.0 mg of aflibercept injection at 4 week intervals through Week 12.
- Aflibercept Injection 2.0mg q12: Participants received 2.0 mg of aflibercept injection at 12 week intervals through Week 12.
- Aflibercept Injection 4.0mg q12: Participants received 4.0 mg of aflibercept injection at 12 week intervals through Week 12.
- Total: Total of all reporting groups
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12 | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 31 | 157
Age Continuous [Mean (Standard Deviation); unit: years] | 79.6 (7.56) [0 to 0] | 78.5 (10.12) [0 to 0] | 74.9 (7.63) [0 to 0] | 79.6 (8.91) [0 to 0] | 78.3 (5.97) [0 to 0] | 78.2 (8.25) [0 to 0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 (0) [0 to 0] | 25 (0) [0 to 0] | 20 (0) [0 to 0] | 16 (0) [0 to 0] | 20 (0) [0 to 0] | 98
  Male | 15 (0) [0 to 0] | 7 (0) [0 to 0] | 11 (0) [0 to 0] | 15 (0) [0 to 0] | 11 (0) [0 to 0] | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 (0) [0 to 0] | 1 (0) [0 to 0] | 2 (0) [0 to 0] | 1 (0) [0 to 0] | 0 (0) [0 to 0] | 4
  Not Hispanic or Latino | 32 (0) [0 to 0] | 31 (0) [0 to 0] | 29 (0) [0 to 0] | 30 (0) [0 to 0] | 31 (0) [0 to 0] | 153
  Unknown or Not Reported | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 1 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 1
  Asian | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0
  Native Hawaiian or Other Pacific Islander | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0
  Black or African American | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0
  White | 32 (0) [0 to 0] | 32 (0) [0 to 0] | 30 (0) [0 to 0] | 31 (0) [0 to 0] | 31 (0) [0 to 0] | 156
  More than one race | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0
  Unknown or Not Reported | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0
Central Retinal/Lesion Thickness (CR/LT) [Mean (Standard Deviation); unit: µm] | 442.2 (109.81) [0 to 0] | 442.6 (136.60) [0 to 0] | 453.3 (143.93) [0 to 0] | 447.0 (119.11) [0 to 0] | 497.5 (191.17) [0 to 0] | 456.4 (142.41) [0 to 0]
Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: letters read] — BCVA as Measured by 4 Meter Early Treatment Diabetic Retinopathy Study (ETDRS)eye charts/measures
  letters read | 54.1 (13.77) [0 to 0] | 55.6 (11.75) [0 to 0] | 57.9 (12.02) [0 to 0] | 57.2 (10.47) [0 to 0] | 53.0 (14.52) [0 to 0] | 55.5 (12.57) [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of CR/LT From Baseline at Week 12
Description: CR/LT measured in micrometers (µm); lower individual values represent better outcomes.
Time Frame: Baseline and at Week 12
Population: Full Analysis Set (FAS) used for analysis, Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12 | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 31 | 157
μm | -153.5 (113.30) [0 to 0] | -75.6 (110.64) [0 to 0] | -169.2 (138.46) [0 to 0] | -56.3 (133.05) [0 to 0] | -139.8 (228.59) [0 to 0] | -118.8 (155.31) [0 to 0]

2. Secondary Outcome: Mean Percent Change of CR/LT From Baseline at Week 12
Description: CR/LT measured in micrometers (µm); a more negative percentage represents a better outcome
Time Frame: Baseline and at Week 12
Population: FAS used for analysis, LOCF
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Aflibercept Injection 0.5mg q4: Participants received 0.5mg of aflibercept injection at 4 week intervals through Week 12.
- Aflibercept Injection 0.5mg q12: Participants received 0.5mg of aflibercept injection at 12 week intervals through Week 12.
- Aflibercept Injection 2.0mg q4: Participants received 2.0mg of aflibercept injection at 4 week intervals through Week 12.
- Aflibercept Injection 2.0mg q12: Participants received 2.0mg of aflibercept injection at 12 week intervals through Week 12.
- Aflibercept Injection 4.0mg q12: Participants received 4.0mg of aflibercept injection at 12 week intervals through Week 12.
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12 | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 31 | 157
percent change | -32.4 (18.92) [0 to 0] | -15.2 (22.52) [0 to 0] | -33.2 (19.56) [0 to 0] | -10.3 (25.49) [0 to 0] | -21.1 (31.56) [0 to 0] | -22.5 (25.41) [0 to 0]

3. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) From Baseline at Week 12
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity of: letter score of 73 to 25 (20/40 to 20/320) in the study eye; a higher score represents better functioning
Time Frame: Baseline and at week 12
Population: FAS used for analysis, LOCF
Measure: Mean (Standard Deviation); unit: letters read
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12 | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 31 | 157
letters read | 8.8 (9.20) [0 to 0] | 3.8 (11.55) [0 to 0] | 8.3 (10.14) [0 to 0] | 5.2 (8.46) [0 to 0] | 2.6 (8.72) [0 to 0] | 5.7 (9.87) [0 to 0]

4. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters of Vision in the ETDRS Letter Score From Baseline at Week 12
Description: as for outcome 3
Time Frame: At Week 12
Population: FAS used for analysis, LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12 | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 31 | 157
percentage of participants | 18.8 (0) [0 to 0] | 21.9 (0) [0 to 0] | 25.8 (0) [0 to 0] | 16.1 (0) [0 to 0] | 9.7 (0) [0 to 0] | 18.5 (0) [0 to 0]

5. Post Hoc Outcome: Mean Change of CR/LT From Baseline at Week 16
Description: CR/LT measured in micrometers (µm); lower individual values represent better outcomes
Time Frame: Baseline and at Week 16
Population: FAS used for analysis, LOCF
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12 | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 31 | 157
µm | -163.3 (108.13) [0 to 0] | -139.6 (126.41) [0 to 0] | -182.7 (146.75) [0 to 0] | -107.4 (112.22) [0 to 0] | -208.6 (202.07) [0 to 0] | -160.2 (145.34) [0 to 0]

6. Post Hoc Outcome: Mean Change in BCVA as Measured by ETDRS From Baseline at Week 16
Description: as for outcome 3
Time Frame: Baseline and at Week 16
Population: FAS used for analysis, LOCF
Measure: Mean (Standard Deviation); unit: letters read
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12 | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 31 | 157
letters read | 9.3 (9.92) [0 to 0] | 5.6 (12.24) [0 to 0] | 10.0 (9.76) [0 to 0] | 4.3 (10.01) [0 to 0] | 3.9 (9.92) [0 to 0] | 6.6 (10.60) [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) considered related to study treatment were followed until resolution or until the event was considered chronic or stable.
Description: Safety was assessed through reported AEs, clinical laboratory test results, vital signs, and ophthalmic examinations
Arm/Group | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12
Serious Adverse Events (participants affected / at risk) | 11 | 5 | 10 | 7 | 2
Other Adverse Events (participants affected / at risk) | 26 | 25 | 27 | 22 | 22
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0/32 | 0/32 | 0/31 | 1/31 | 0/31
BRAIN NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/32 | 1/32 | 0/31 | 0/31 | 0/31
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/32 | 1/32 | 0/31 | 0/31 | 0/31
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/32 | 0/32 | 0/31 | 1/31 | 0/31
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/32 | 0/32 | 0/31 | 1/31 | 0/31
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/32 | 0/32 | 0/31 | 1/31 | 0/31
DEEP VEIN THROMBOSIS (Vascular disorders) | 0/32 | 1/32 | 0/31 | 0/31 | 0/31
DYSKINESIA OESOPHAGEAL (Gastrointestinal disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
VOLVULUS (Gastrointestinal disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
ASTHENIA (General disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
NON-CARDIAC CHEST PAIN (General disorders) | 0/32 | 1/32 | 0/31 | 0/31 | 0/31
ANGINA PECTORIS (Cardiac disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
ATRIAL FIBRILLATION (Cardiac disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 1/31
BRADYCARDIA (Cardiac disorders) | 0/32 | 0/32 | 0/31 | 0/31 | 1/31
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1/32 | 0/32 | 2/31 | 0/31 | 0/31
CORONARY ARTERY DISEASE (Cardiac disorders) | 0/32 | 0/32 | 2/31 | 0/31 | 0/31
BRONCHITIS (Infections and infestations) | 0/32 | 0/32 | 1/31 | 1/31 | 0/31
CELLULITIS (Infections and infestations) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
GASTROENTERITIS (Infections and infestations) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
PNEUMONIA (Infections and infestations) | 2/32 | 0/32 | 2/31 | 0/31 | 0/31
URINARY TRACT INFECTION (Infections and infestations) | 0/32 | 0/32 | 1/31 | 1/31 | 0/31
FALL (Injury, poisoning and procedural complications) | 1/32 | 0/32 | 1/31 | 0/31 | 0/31
HIP FRACTURE (Injury, poisoning and procedural complications) | 0/32 | 1/32 | 1/31 | 0/31 | 0/31
SKIN LACERATION (Injury, poisoning and procedural complications) | 0/32 | 0/32 | 0/31 | 1/31 | 0/31
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
RENAL FAILURE (Renal and urinary disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
STRESS INCONTINENCE (Renal and urinary disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
URINARY RETENTION (Renal and urinary disorders) | 0/32 | 1/32 | 0/31 | 0/31 | 0/31
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
COORDINATION ABNORMAL (Nervous system disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
DYSARTHRIA (Nervous system disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
SPINAL CORD DISORDER (Nervous system disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
PILONIDAL SINUS REPAIR (Surgical and medical procedures) | 0/32 | 1/32 | 0/31 | 0/31 | 0/31
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0/32 | 0/32 | 1/31 | 0/31 | 0/31
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0/32 | 0/32 | 0/31 | 1/31 | 0/31
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0/32 | 0/32 | 0/31 | 0/31 | 1/31
RETINAL DETACHMENT (Eye disorders) | 0/32 | 1/32 | 0/31 | 0/31 | 0/31 — Fellow Eye
VISUAL ACUITY REDUCED (Eye disorders) | 0/32 | 0/32 | 0/31 | 0/31 | 0/31 — Fellow Eye
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0/32 | 0/32 | 0/31 | 0/31 | 1/31 — Fellow Eye
UVEITIS (Eye disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 0/31 — Study Eye
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Aflibercept Injection 0.5mg q4 | Aflibercept Injection 0.5mg q12 | Aflibercept Injection 2.0mg q4 | Aflibercept Injection 2.0mg q12 | Aflibercept Injection 4.0mg q12
ANAEMIA (Blood and lymphatic system disorders) | 0/32 | 1/32 | 3/31 | 0/31 | 0/31
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1/32 | 0/32 | 2/31 | 0/31 | 0/31
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0/32 | 0/32 | 2/31 | 0/31 | 1/31
HYPERTENSION (Vascular disorders) | 6/32 | 1/32 | 2/31 | 0/31 | 3/31
HYPOTENSION (Vascular disorders) | 0/32 | 0/32 | 2/31 | 0/31 | 0/31
CONSTIPATION (Gastrointestinal disorders) | 5/32 | 1/32 | 0/31 | 0/31 | 1/31
DIARRHOEA (Gastrointestinal disorders) | 1/32 | 1/32 | 0/31 | 1/31 | 2/31
FLATULENCE (Gastrointestinal disorders) | 0/32 | 2/32 | 0/31 | 0/31 | 0/31
NAUSEA (Gastrointestinal disorders) | 3/32 | 0/32 | 0/31 | 1/31 | 1/31
CHEST PAIN (General disorders) | 2/32 | 0/32 | 0/31 | 0/31 | 0/31
ANGINA PECTORIS (Cardiac disorders) | 2/32 | 0/32 | 1/31 | 1/31 | 0/31
BRADYCARDIA (Cardiac disorders) | 1/32 | 0/32 | 2/31 | 0/31 | 0/31
SEASONAL ALLERGY (Immune system disorders) | 4/32 | 2/32 | 0/31 | 0/31 | 1/31
BRONCHITIS (Infections and infestations) | 5/32 | 2/32 | 1/31 | 1/31 | 3/31
CELLULITIS (Infections and infestations) | 0/32 | 0/32 | 0/31 | 2/31 | 1/31
CYSTITIS (Infections and infestations) | 2/32 | 0/32 | 1/31 | 1/31 | 0/31
GASTROENTERITIS VIRAL (Infections and infestations) | 0/32 | 0/32 | 2/31 | 0/31 | 1/31
HERPES ZOSTER (Infections and infestations) | 0/32 | 2/32 | 0/31 | 0/31 | 0/31
INFLUENZA (Infections and infestations) | 0/32 | 2/32 | 2/31 | 0/31 | 2/31
NASOPHARYNGITIS (Infections and infestations) | 3/32 | 1/32 | 3/31 | 1/31 | 2/31
PNEUMONIA (Infections and infestations) | 3/32 | 0/32 | 2/31 | 1/31 | 1/31
RHINOVIRUS INFECTION (Infections and infestations) | 0/32 | 0/32 | 2/31 | 0/31 | 0/31
SINUSITIS (Infections and infestations) | 2/32 | 1/32 | 2/31 | 1/31 | 3/31
TOOTH ABSCESS (Infections and infestations) | 1/32 | 1/32 | 1/31 | 2/31 | 0/31
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3/32 | 1/32 | 2/31 | 6/31 | 3/31
URINARY TRACT INFECTION (Infections and infestations) | 1/32 | 3/32 | 6/31 | 1/31 | 2/31
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0/32 | 1/32 | 0/31 | 2/31 | 1/31
FALL (Injury, poisoning and procedural complications) | 2/32 | 1/32 | 1/31 | 0/31 | 0/31
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0/32 | 0/32 | 0/31 | 0/31 | 2/31
BLOOD CREATININE INCREASED (Investigations) | 0/32 | 1/32 | 0/31 | 2/31 | 1/31
BLOOD GLUCOSE INCREASED (Investigations) | 0/32 | 2/32 | 1/31 | 1/31 | 0/31
BLOOD UREA INCREASED (Investigations) | 0/32 | 1/32 | 0/31 | 2/31 | 0/31
DEHYDRATION (Metabolism and nutrition disorders) | 1/32 | 1/32 | 2/31 | 0/31 | 1/31
GOUT (Metabolism and nutrition disorders) | 1/32 | 2/32 | 0/31 | 0/31 | 0/31
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 4/32 | 0/32 | 0/31 | 0/31 | 0/31
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0/32 | 2/32 | 0/31 | 0/31 | 0/31
DIZZINESS (Nervous system disorders) | 1/32 | 0/32 | 2/31 | 1/31 | 0/31
HEADACHE (Nervous system disorders) | 1/32 | 3/32 | 1/31 | 0/31 | 1/31
SINUS HEADACHE (Nervous system disorders) | 1/32 | 2/32 | 2/31 | 0/31 | 2/31
ANXIETY (Psychiatric disorders) | 0/32 | 0/32 | 2/31 | 0/31 | 0/31
DEPRESSION (Psychiatric disorders) | 0/32 | 1/32 | 2/31 | 0/31 | 0/31
INSOMNIA (Psychiatric disorders) | 2/32 | 0/32 | 1/31 | 0/31 | 0/31
COUGH (Respiratory, thoracic and mediastinal disorders) | 2/32 | 1/32 | 2/31 | 1/31 | 2/31
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2/32 | 0/32 | 1/31 | 2/31 | 0/31
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1/32 | 0/32 | 0/31 | 0/31 | 2/31
RASH (Skin and subcutaneous tissue disorders) | 2/32 | 0/32 | 1/31 | 0/31 | 1/31
BLEPHARITIS (Eye disorders) | 2/32 | 0/32 | 2/31 | 3/31 | 1/31 — Fellow Eye
CATARACT (Eye disorders) | 0/32 | 1/32 | 1/31 | 1/31 | 2/31 — Fellow Eye
CATARACT NUCLEAR (Eye disorders) | 3/32 | 0/32 | 2/31 | 1/31 | 0/31 — Fellow Eye
CATARACT SUBCAPSULAR (Eye disorders) | 0/32 | 2/32 | 0/31 | 1/31 | 2/31 — Fellow Eye
CHOROIDAL NEOVASCULARISATION (Eye disorders) | 0/32 | 1/32 | 2/31 | 1/31 | 0/31 — Fellow Eye
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 2/32 | 0/32 | 2/31 | 2/31 | 1/31 — Fellow Eye
DETACHMENT OF RETINAL PIGMENT EPITHELIUM (Eye disorders) | 2/32 | 1/32 | 0/31 | 0/31 | 1/31 — Fellow Eye
DRY EYE (Eye disorders) | 1/32 | 0/32 | 1/31 | 2/31 | 0/31 — Fellow Eye
LACRIMATION INCREASED (Eye disorders) | 0/32 | 0/32 | 0/31 | 0/31 | 2/31 — Fellow Eye
REFRACTION DISORDER (Eye disorders) | 1/32 | 4/32 | 1/31 | 1/31 | 3/31 — Fellow Eye
RETINAL HAEMORRHAGE (Eye disorders) | 0/32 | 2/32 | 1/31 | 3/31 | 0/31 — Fellow Eye
RETINAL OEDEMA (Eye disorders) | 1/32 | 2/32 | 1/31 | 0/31 | 0/31 — Fellow Eye
RETINAL PIGMENT EPITHELIOPATHY (Eye disorders) | 2/32 | 3/32 | 0/31 | 1/31 | 1/31 — Fellow Eye
VISUAL ACUITY REDUCED (Eye disorders) | 1/32 | 1/32 | 4/31 | 1/31 | 1/31 — Fellow Eye
VITREOUS DETACHMENT (Eye disorders) | 4/32 | 1/32 | 2/31 | 3/31 | 4/31 — Fellow Eye
VITREOUS FLOATERS (Eye disorders) | 2/32 | 0/32 | 0/31 | 1/31 | 1/31 — Fellow Eye
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1/32 | 3/32 | 3/31 | 2/31 | 1/31 — Fellow Eye
EYE INFLAMMATION (Eye disorders) | 2/32 | 0/32 | 0/31 | 1/31 | 1/31 — Study Eye
EYE IRRITATION (Eye disorders) | 5/32 | 0/32 | 1/31 | 0/31 | 1/31 — Study Eye
EYE PAIN (Eye disorders) | 5/32 | 2/32 | 4/31 | 1/31 | 3/31 — Study Eye
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 3/32 | 0/32 | 1/31 | 0/31 | 0/31 — Study Eye
LACRIMATION DECREASED (Eye disorders) | 0/32 | 0/32 | 0/31 | 0/31 | 2/31 — Study Eye
MACULAR DEGENERATION (Eye disorders) | 0/32 | 0/32 | 0/31 | 0/31 | 2/31 — Study Eye
MACULOPATHY (Eye disorders) | 1/32 | 0/32 | 0/31 | 2/31 | 1/31 — Study Eye
PHOTOPSIA (Eye disorders) | 1/32 | 0/32 | 0/31 | 2/31 | 3/31 — Study Eye
PUNCTATE KERATITIS (Eye disorders) | 0/32 | 0/32 | 1/31 | 2/31 | 2/31 — Study Eye
RETINAL DEPIGMENTATION (Eye disorders) | 2/32 | 0/32 | 0/31 | 0/31 | 0/31 — Study Eye
SUBRETINAL FIBROSIS (Eye disorders) | 2/32 | 1/32 | 1/31 | 2/31 | 2/31 — Study Eye
VISION BLURRED (Eye disorders) | 2/32 | 0/32 | 0/31 | 0/31 | 1/31 — Study Eye
VISUAL DISTURBANCE (Eye disorders) | 2/32 | 1/32 | 0/31 | 2/31 | 3/31 — Study Eye

LIMITATIONS AND CAVEATS:
This is a phase 2 study with small numbers of patients per group limiting the conclusions that can be drawn from the resulting data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the trial, the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review; provided that the sponsor can remove confidential or proprietary information from such communications. The sponsor cannot require other changes to the communication and cannot extend the embargo.